CLINICAL TRIAL: NCT04837612
Title: Observational Study for Patients With Dilated Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Cheng Huang, PROFESSOR, Guangdong Provincial People's Hospital
Other Study IDs: GDREC2019546HR1
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: DCM - Dilated Cardiomyopathy
Keywords: all-cause mortality; cardiovascular death; hospitalization for heart failure; heart transplatation
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, whole blood, and white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with dilated cardiomyopathy: Subjects diagnosed with dilated cardiomyopathy by medical history, physical examination and echocardiography.
  Interventions: Other: No intervention nor exposure

INTERVENTIONS:
Other: No intervention nor exposure — As an observational study, no intervention nor exposure is interested.

SUMMARY:
Observational study on patients with dilated cardiomyopathy aims to investigate the correlation between cardiac fibrosis, as indicated by cardiac magnetic resonance, and the prognosis of patients with dilated cardiomyopathy, and further to explore biomarkers for cardiac fibrosis and adverse prognosis of dilated cardiomyopathy. Therefore, endpoints indluding all-cause mortality, cardiovascular death, ventricular arrythmia, non-fatal stroke, non-fatal myocardial infarction, sudden death, successful cardiopulmonary resuscitation will be evaluated.

DETAILED DESCRIPTION:
In this observational study on patients with dilated cardiomyopathy, 500 eligible patients, who were diagnosed as dilated cardiomyopathy by echocardiography, will be recruited with a median follow up of 5 years.Patients will be excluded who develop cardiac enlargement caused by other factors such as myocardial ischemia, myocarditis, diabetic cardiomyopathy, valvular heart disease, congenital heart disease; who had underwent heart transplatation; who are not suitable for the present study due to maligant tumor or severe trauma.

Eligible individuals, identified based on echocardiography and medical records, were invited to a community clinic by phone. For eligible individuals, study data were comprised of a self-administered questionnaire, anthropometric features, laboratory examinations, echocardiographic and/or cardiac magetic resnonance data. Anthropometric data were measured by experienced research staff in the morning under standardized conditions. Echocardiographic measuring were performed by three skilled sonographers independently, based on routine protocols on an HP5500 (Phillips Medical System, Boston, Massachusetts, USA) per current guidelines. Venous blood samples were collected in the morning following overnight fasting. Laboratory procedures were performed under standardized conditions.

Endpoints including all-cause mortality, cardiovascular death, sudden death (ICD-Code I46.1, R96), ventricular tachycardia(ICD-code I47.2)/fibrillation/flutter(ICD-code I49.0), hospitalization for heart failure(ICD-Code I50), heart transplatation ((ICD-Code Z94.1), non-fatal stroke(ICD-Code I60, I61, I63, I64), non-fatal myocardial infarction (ICD-Code I21), sudden death (ICD-Code I46.1, R96), successful cardiopulmonary resuscitation (ICD-Code I46.0) will be evaulated.

Across the whole observational study, 50 endpoints are anticipated to occur annually, and therefore the sample size was estimated to be approximately 500 subjects.

Data collection and management will be conducted via electronic data collection (EDC). Source data will be checked regularly to assess the accuracy and completeness. For statistical analysis, continuous variables are presented as mean±standard deviation (SD), and compared by the Student t-test. Categorical variables are presented as frequency and assessed by the χ2 test. SAS 9.4 for Windows (release 6.11, USA) is to be utilized for statistical analysis.

ELIGIBILITY:
Inclusion Criteria: Dilated cardiomyopathy diagnosed by medical history, physical examination and echocardiography.

-

Exclusion Criteria:

* Cardiac enlargement caused by other factors such as myocardial ischemia, myocarditis, diabetic cardiomyopathy, valvular heart disease, congenital heart disease, Patients who had underwent heart transplatation. Individuals not suitable for the present study due to maligant tumor or severe trauma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with dilated cardiomyopathy by medical history, physical examination and echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 5 YEARS.
  All-cause mortality refers to death from any causes.

SECONDARY OUTCOMES:
Cardiovascular death | 5 YEARS.
  Cardiovascular death include death caused by stroke, MI, HF, sudden death or any other death attributed to cardiovascular diseases.
Ventricular tachycardia and fibrillation and flutter | 5 YEARS.
  Ventricular tachycardia is an abnormally fast heart beat (with three or more consecutive heart beats at least 100 beats per minute) that originates from one of the ventricles in the heart (ICD-code I47.2), respectively.Ventricular fibrillation (VF) is a very rapid (150-500 bpm) irregularly irregular disorganized ventricular rhythm of varying configuration; with time, the amplitude of the fibrillation wave becomes progressively smaller, particularly immediately before death. Ventricular flutter (VFL) is a very rapid (180-250 bpm) and regular ectopic ventricular rhythm with undulations of equal amplitude and usually rapidly degenerates to VF(ICD-code I49.0).
nonfatal stroke | 5 YEARS.
  Stroke (ICD-Code I60, I61, I63, I64) is a focal neurological deficit with symptoms continuing for more than 24 hours or leading to death with no apparent cause other than vascular. Stroke as an endpoint in this study includes definite ischemic stroke, primary intracerebral hemorrhage and subarachnoid hemorrhage with evidence from CT or MRI scan within 14 days of onset or autopsy confirmation, and stroke of unknown type etiology when CT, MRI, or autopsy are not done and information is inadequate to diagnose the etiology definitely.
nonfatal myocardial infarction | 5 YEARS.
  Acute myocardial infarction (MI) (ICD-Code I21) is defined when any one of the following criteria occurs. (1) Detection of a rise and/or fall of cardiac biomarker values, with at least one value above the 99th percentile upper reference limit and with at least one of the following manifestations: symptoms of ischaemia that should have lasted for at least 30 minutes and should not have been responsive to sublingual administration of nitrates; new or presumed new significant ST-segment-T wave changes or new left bundle branch block (LBBB); development of pathological Q waves in the ECG; imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. (2) Identification of an intracoronary thrombus by angiography or autopsy. (3) Cardiac death with symptoms suggestive of myocardial ischaemia and presumed new ischaemic ECG changes or new LBBB, but death occurred before cardiac biomarkers were obtained, or before cardiac biomarker values would be increased.
sudden death | 5 YEARS.
  Sudden death (ICD-Code I46.1, R96) encompasses any death of unknown origin occurring instantly or within an estimated 24 hours after the onset of acute symptoms as well as unattended death for which no likely cause can be established by autopsy or recent medical history.
Cardiac arrest with successful resuscitation | 5 YEARS.
  ICD-Code I46.0
Hospitalization for heart failure | 5 YEARS
  Congestive heart failure (HF) (ICD-Code I50) requires the presence of three conditions, namely symptoms, such as dyspnea, clinical signs, such as ankle edema or crepitations, and the necessity to initiate treatment with open-label diuretics, vasodilators or antihypertensive drugs. HF cases may also be adjudicated as chronic stable HF but this is not considered an outcome of the present study.
Heart transplatation | 5 YEARS
  Heart replaced by heterogenous or homogenoustransplant due to end-stage heart failure. (ICD-Code Z94.1).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Huang, PhD, Principal Investigator — Guangdong Cardiovascular institute, Dongchuan Road,96#, Guangzhou City, Guangdong Province
Locations (1):
- Guangdong cardiovascular institute, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
A part of participants do not want their privacy to be shared by other reserchers.